CLINICAL TRIAL: NCT07253376
Title: Validity and Reliability Analysis of the Turkish Version of The Parkinson Disease Cognitive Functional Rating Scale
Brief Title: Turkish Validation of the Parkinson Disease Cognitive Functional Rating Scale
Status: Enrolling by invitation | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: T.C. Sağlık Bakanlığı Ankara Bilkent Şehir Hastanesi (Other)
Responsible Party: Principal Investigator, Arzu Güçlü Gündüz, Professor, PhD, PT, Gazi University
Other Study IDs: TABED 1-25-1618
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cognition; Parkinson's Disease; Reliability and Validity; Cognitive Functions; Cognitive Functioning
Keywords: Parkinson's disease; Cognition; Cognitive Functions; Reliability; Validity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with Parkinson's Disease: Participants diagnosed with Parkinson's disease who will complete the Turkish version of the Parkinson's Disease-Cognitive Functional Rating Scale (PD-CFRS) for validity and reliability analysis.

SUMMARY:
The aim of the present study is to translate the Parkinson's Disease-Cognitive Functional Rating Scale into Turkish (PD-CFRS-Turkish version) and to evaluate its validity and reliability.

DETAILED DESCRIPTION:
The Parkinson's Disease-Cognitive Functional Rating Scale (PD-CFRS) is one of the Parkinson's disease-specific instruments developed to assess a broad range of functional impairments resulting from cognitive deficits in individuals with Parkinson's disease (PD). The PD-CFRS is specifically designed to evaluate cognitive dysfunction while minimizing the confounding effects of motor symptoms.

The scale consists of 12 items that assess whether the patient experiences difficulties in performing activities such as managing money and household finances, arranging vacations or meetings, handling personal correspondence, checking medication schedules, organizing daily routines, using electrical appliances, understanding public transportation, dealing with unforeseen situations, expressing intentions, comprehending written information, and using a mobile phone.

Each item is rated on a 3-point scale ranging from 0 to 2. If the participant has never performed the activity in question, a score of 8 is assigned. At the end of the assessment, the average score for items rated between 0 and 2 is calculated and rounded to the nearest whole number. This value replaces all items initially scored as 8. Once all substituted scores are assigned, the total score is obtained by summing all item scores. The administration time for the scale is approximately 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with idiopathic Parkinson's disease by a neurologist.
* Evaluated between Stage 1-3 according to the Hoehn and Yahr Staging Scale.
* Aged 40 years or older.
* Agreed to participate in the study after being given sufficient information.

Exclusion Criteria:

* Patients with a Montreal Cognitive Assessment score of 20 and below.
* Patients with cardiovascular, vestibular, musculoskeletal or additional neurological disease.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study has a multicenter design. The participating sites are as follows:
  Ankara Bilkent City Hospital, Physical Therapy and Rehabilitation Hospital- designated as Site 1. Participants at this site will include individuals diagnosed with Parkinson's disease (PD) who are currently receiving treatment at the hospital and have consented to participate in the study.
  Gazi University, Faculty of Health Sciences, Neurological Physical Therapy and Rehabilitation Unit - designated as Site 2. Participants at this site will include individuals diagnosed with PD who have been referred to the unit and have consented to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Validity of the Turkish Version of the Parkinson's Disease Cognitive Functional Rating Scale (PD-CFRS) | Single assessment.
  The original English version of the PD-CFRS, developed by the Movement Disorders community (Barcelona, Spain), assesses the functional impact of cognitive impairment in individuals with Parkinson's disease.
  The validity of the PD-CFRS Turkish version will be evaluated through convergent and discriminant construct analyses. Convergent validity will be assessed by examining partial Pearson correlations between PD-CFRS scores and MMSE and MoCA scores, controlling for age at onset, education level, and disease duration. Discriminant validity will be analyzed using binary logistic regression with MMSE and MoCA scores and disease duration as independent variables.

SECONDARY OUTCOMES:
Reliability of the Turkish Version of the Parkinson's Disease Cognitive Functional Rating Scale (PD-CFRS) | Repeated measurements will be conducted at a 2 week interval.
  Test-retest reliability will be assessed by repeating the PD-CFRS administration after a two-week interval by the same examiner. The scale evaluates participants' cognitive skills over the previous two weeks. Reliability will be calculated using the Intraclass Correlation Coefficient (ICC).
Mini Mental State Examination (MMSE) Score | Single assessment.
  Assessment of general cognitive function, including attention, orientation, memory, verbal responses, following verbal and written commands, sentence writing, and copying complex figures. Scores <24 indicate cognitive impairment. The score obtained from the test will be recorded.
Montreal Cognitive Assessment (MoCA) Score | Single assessment.
  Montreal Cognitive Assessment (MoCA), which provides a general cognitive screening in different cognitive functions such as attention, concentration, executive functions, memory, language, visual structuring skills, abstract thought, calculation and orientation, will be used in the general evaluation of cognition. MoCA is an effective scale especially in the evaluation of mild cognitive impairments in Parkinson's disease (PD). The cut-off score range of MoCA has been shown to be 18-26 points in individuals with PD who has mild cognitive impairment. The administration of MoCA takes approximately 10 minutes. The highest total score that can be obtained from the test is 30. Accordingly, a score of 21 points and above is considered normal. The score obtained from the test will be recorded.
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3: Motor Examination Score | Single assessment.
  Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) consists of 4 parts, like the classic UPDRS. The severity of the patients' motor symptoms will be assessed using the Motor Examination part, which is the 3rd part of the MDS-UPDRS. MDS-UPDRS Part 3 consists of 18 items. All items in the scale are scored between 0 (Normal) and 4 (Severe) points. The score obtained from the test will be recorded.
Hoehn and Yahr Scale | Single assessment.
  Short staging system to evaluate the severity of Parkinson's disease symptoms.
Hospital Anxiety and Depression Scale (HADS) Scores | Single assessment.
  Assessment of anxiety (HADS-A) and depression (HADS-D) symptoms. The fourteen-item HADS includes a mixed seven-item Anxiety subscale (HADS-A) and a Depression subscale (HADS-D). Each item is scored from a four-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Adıgüzel, Prof., MD., Study Director — Ankara City Hospital Bilkent; Arzu Güçlü Gündüz, Prof., PT., Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Faculty of Health Sciences, Ankara
  - Ankara Bilkent City Hospital, Physical Medicine and Rehabilitation Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Ozdilek B, Kenangil G. Validation of the Turkish Version of the Montreal Cognitive Assessment Scale (MoCA-TR) in patients with Parkinson's disease. Clin Neuropsychol. 2014;28(2):333-43. doi: 10.1080/13854046.2014.881554. Epub 2014 Feb 17. PMID 24528299
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Kulisevsky J, Fernandez de Bobadilla R, Pagonabarraga J, Martinez-Horta S, Campolongo A, Garcia-Sanchez C, Pascual-Sedano B, Ribosa-Nogue R, Villa-Bonomo C. Measuring functional impact of cognitive impairment: validation of the Parkinson's disease cognitive functional rating scale. Parkinsonism Relat Disord. 2013 Sep;19(9):812-7. doi: 10.1016/j.parkreldis.2013.05.007. Epub 2013 Jun 15. PMID 23773412
- [Background] Kline, P. (1994). An Easy Guide to Factor Analysis (1st ed.). Routledge.
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Kawabe H, Nagano H. [Case of sarcoidosis with marked changes at the site of Progynon depot injection of 4 years duration]. Saishin Igaku. 1969 Dec;24(12):2595-8. No abstract available. Japanese. PMID 5363424
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252